CLINICAL TRIAL: NCT05052398
Title: Proof of Principle Study Evaluating the Effects of Gonyautoxins, Paralytic Shellfish Poisoning (PSP) NEURO SERUM, on Objective and Subjective Symptoms of Chemotherapy-induced Peripheral Neuropathy (CINP)
Brief Title: Proof of Principle Study Evaluating Gonyautoxins NEURO SERUM, on Chemotherapy-induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Algenis SpA (Industry)
Collaborators: Oncoclínicas (Industry)
Responsible Party: Principal Investigator, Mariane Sousa Fontes Dias, Principal Investigator, Oncoclínicas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Onco-2020
Record Dates: First submitted 2021-08-10; First posted 2021-09-22 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: Part 1 is a 2-stage, 2-cohort, open-label study where up to 38 pts with G>2 CIPN secondary to taxanes and other anti-neoplastic drugs will receive PSP NEURO SERUM (PNS) thrice a day for 28 days. Twelve patients will be evaluated in stage 1, expecting a 20% response per cohort to proceed to stage 2. If needed 7 patients will be recruited, expecting 4/19 response in each cohort. If the number of responses is not met, recruitment will be halted. Part 2 consists of 2 randomized groups of 26 patients each, one control and one experimental group. The population will follow an adaptive approach, considering which cohorts benefited the most from the effects of PNS in Part 1. The 52 patients will be allocated in a 1:1 ratio to Arm A (control) or Arm B with the objective of estimating and comparing the responses of tactile sensitivity using the Semmes-Weinstein monofilament test in hands. Arm A will receive placebo 3 times/day for 28 days, and Arm B will receive PNS 3 times/day for 28 days.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSP NEURO SERUM (Active Comparator): Active arm in which 26 patients will receive PSP NEURO SERUM in their hands three times a day for 28 days. Each application will consist of 1 g of PSP NEURO SERUM.
  Interventions: Drug: PSP NEURO SERUM
- Placebo of PSP NEURO SERUM (Placebo Comparator): Placebo arm in which 26 patients will receive Placebo PSP NEURO SERUM (same ingredients as PSP NEURO SERUM except for the active ingredient that is replace with water) in their hands three times a day for 28 days. Each application will consist of 1 g of Placebo PSP NEURO SERUM.
  Interventions: Drug: Placebo PSP NEURO SERUM

INTERVENTIONS:
Drug: PSP NEURO SERUM — PSP NEURO SERUM is a topical product that contains a concentration of Paralytic Shellfish Toxins of 10 micrograms/mL of equivalent of Gonyautoxin 2/3. Each patient will apply 1 g of PSP NEURO SERUM in their hands, three times a day.
  Arms: PSP NEURO SERUM
Drug: Placebo PSP NEURO SERUM — Placebo PSP NEURO SERUM is the same topical product as PSP NEURO SERUM without the active ingredient. Each patient will apply 1 g of Placebo PSP NEURO SERUM in their hands, three times a day.
  Arms: Placebo of PSP NEURO SERUM

SUMMARY:
Proof-of-concept study to assess the effects of gonyautoxins (PSP NEURO SERUM) on safety and tactile sensitivity on patients with chemotherapy-induced peripheral neuropathy (CIPN). This is a multicenter, prospective proof-of-concept study in patients with solid tumors affected by CIPN. The study will be divided into two parts: Part 1 will assess the activity and tolerability of PSP NEURO SERUM and part 2 consists of a randomized cohort that will compare the activity of PSP NEURO SERUM vs placebo. Part 2 will depend on the results of part 1. If there are less than 8 responses in part 1, the study will be interrupted, and it will not be recommended to proceed with part 2.

DETAILED DESCRIPTION:
A multicenter, prospective proof-of-concept study in patients with solid tumors who developed chemotherapy-induced peripheral neuropathy (CIPN) in upper limbs, equal or greater than grade 2, according to NCI-CTCAE version 5.0. Patients must have been treated with cytotoxic agents known to cause CIPN in neoadjuvant, adjuvant or palliative setting. The primary objective is to assess the effects of gonyautoxins (PSP NEURO SERUM) on tactile sensitivity and safety on patients with CIPN. The study will be divided into two parts, 1 and 2 and the investigational treatment will have a maximum duration of 4 weeks (28 days).

Part 1 is a two-stage (stage 1 and stage 2), two-cohort (C1 and C2), open-label study where up to 38 pts with G>2 CIPN secondary to taxanes (C1) and other anti-neoplastic drugs (C2) will receive PSP NEURO SERUM thrice a day for 28 days. Twelve patients will be evaluated in stage 1, expecting a 20% response (2/12) in each cohort to proceed to stage 2. If needed, additional 7 patients will be recruited to stage, expecting 4/19 response in each cohort. If the number of responses is not met in a specific cohort, recruitment will be halted. The transition to the randomized part 2 will be determined by the efficacy in part 1 (stratified analysis of C1 and C2 or overall population).

The primary objective of Part 1 is to evaluate response of the tactile sensation as assessed by the Semmes-Weinstein monofilament test and to evaluate safety and toxicity (type, frequency, grade and causality of adverse effects) of PSP NEURO SERUM according to NCI-CTCAE v5.0.

The secondary objectives of Part 1 are to:

1. Evaluate the improvement of overall neurological examination as assessed by the clinical version of Total Neuropathy Score (TNSc)
2. Evaluate the improvement of manipulative dexterity and agility as assessed by the nine-hole pegboard test (NHPT).
3. Evaluate the improvement in patient reported symptoms as assessed by the Patient Neuropathy Questionnaire (PNQ).
4. Evaluate the improvement of quality of life by using the Portuguese version of the 30-item European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC Quality of Life Questionnaire (QLQ-C30)) version.

A patient will have responded to the CIPN in the study if there is a documented improvement of 30% (two sizes of evaluator) and / or normalization of the baseline pretreatment assessment as assessed by the Semmes-Weinstein monofilament test. A patient will have progressed CIPN in the study if there is a documented worsening in tactile sensation assessed by the Semmes-Weinstein monofilament test. Worse tactile sensation is defined as the change in one (1) size of the monofilament evaluator.

Part 2 of the study consists of two randomized groups of 26 patients each, one control group, and one experimental group, resulting in a total of 52 patients. The composition of the study population will follow an adaptive approach, considering which cohorts benefited the most from the effects of PSP NEURO SERUM in Part 1. Due to the greater benefit observed in cohort 1, we will proceed in Part 2 with only the population of patients who developed peripheral neuropathy secondary to taxanes.

The 52 patients will be allocated in a 1:1 ratio to either Arm A (control, n=26) or Arm B (experimental, n=26) with the objective of estimating and comparing the responses of tactile sensitivity using the Semmes-Weinstein monofilament test in hands caused by NPIQ. Patients in Arm A will receive a placebo (topical formulation composed of the same excipients without the active ingredient) three times a day for 28 days, and patients in Arm B will receive PSP NEURO SERUM (topical formulation) three times a day for 28 days.

This study will follow a two-stage randomized analysis approach with the expectation that the control group will have up to 20% response rate compared to 50% in the experimental group. An independent committee will assess and monitor the data collection results, allowing or disallowing the continuation of the analysis. The first stage will occur when both groups reach 50% of patients with complete validation, where a partial evaluation of necessary criteria will take place to proceed with data collection until reaching the required sample size for the final analysis (second stage).

In Part 2, patients with symptoms in their feet will be offered the possibility of using PSP NEURO SERUM/placebo on their lower limbs. The evaluation of symptoms will be assessed by extrapolation based on data collected by the EORTC QLQ CIPN20 Neuropathy Questionnaire.

The primary objective of Part 2 is to Evaluate tactile sensitivity response through the monofilament test of Semmes-Weinstein.

The secondary objectives of Part 2 are to:

1. Evaluate the improvement of overall neurological examination as assessed by the clinical version of Total Neuropathy Score (TNSc)
2. Evaluate the improvement of manipulative dexterity and agility as assessed by the nine-hole pegboard test (NHPT).
3. Evaluate the improvement in patient reported symptoms as assessed by the Patient Neuropathy Questionnaire (PNQ).EORTC CIPN20
4. Assess safety and toxicity as per NCI-CTCAE v5.0 (National Cancer Institute - Common Toxicity Criteria For Adverse Events). Adverse events will be collected weekly and at the visit of safet/monitoring;
5. Evaluate the improvement of quality of life by using the Portuguese version of the 30-item European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC Quality of Life Questionnaire (QLQ-C30)) version.

The study procedures include:

1. Screening Assessments (Part 1 and 2)
2. Pre-treatment / Baseline Assessments (D1) (Part 1 and 2)
3. D7 (± 1 day) - Assessments during Treatment (Part 1)
4. D14 (± 1 day) - Assessments during Treatment (Part 1 and 2)
5. D21 (± 1 day) - Assessments during Treatment (Part 1)
6. End of Treatment (D28 + 3 days) (Part 1 and 2)
7. Safety Follow-up Visit (30 ± 7 days from the last dose) (Part 1 and 2)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥18 years
3. Histological diagnosis of cancer (hematologic or solid tumors).
4. Part 1: Treatment with antineoplastic agents that induce peripheral neuropathy in neoadjuvant, adjuvant, or metastatic scenario; Part 2: Treatment with taxanes peripheral neuropathy inducers in the neoadjuvant, adjuvant, or metastatic scenario.
5. Peripheral sensory neuropathy grade 2 or higher on upper limbs as per NCI-CTCAE v5.0. and with alteration of the Semmes Weinstein monofilament test.
6. Part 1: Diagnosis of peripheral sensory neuropathy during treatment with antineoplastic agents drugs that induce peripheral neuropathy or up to 2 weeks after the last chemotherapy infusion; Part 2: Diagnosis of peripheral sensory neuropathy during treatment with peripheral neuropathy-inducing taxanes or up to 2 weeks after last chemotherapy infusion.
7. Part 1: Patients with chronic symptoms related to peripheral sensory neuropathy who have completed treatment with peripheral neuropathy-inducing antineoplastic agents for more than 2 weeks and without any exclusion criteria, may be included. Part 2: Patients with chronic symptoms related to sensory peripheral neuropathy who completed treatment with peripheral neuropathy-inducing taxanes for more than 2 weeks and no exclusion criteria, can be included.
8. Patients using neuropathic pain modulators will be allowed if there is no dose adjustments in the last 2 weeks and if sensory symptoms persist related to CIPN, or if the use is for another indication.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
10. Documented willingness to use an effective contraceptive method while participate in the study for male patients with partners or female participants with the potential to become pregnant.
11. Part 1: Hand skin and cuticles must be intact. Part 2: Skin of hands, feet and cuticles must be intact.

Exclusion Criteria:

1. Prior treatment with gonyautoxins or any small molecule neurotoxins.
2. Female participants who are pregnant (positive urine pregnancy test), who have an infant they are breastfeeding, or intend to become pregnant within 3 months.
3. History of peripheral sensory neuropathy attributed to any cause other than chemotherapy.
4. Patients receiving systemic treatment that has among its common side effects (> 1%) peripheral neuropathy, or who have received the same within the last 2 weeks. The use during the study of systemic drugs such as hormone therapy (e.g. tamoxifen, aromatase inhibitor, etc), or other agents that do not have among their common side effects (>1%) peripheral neuropathy, will be allowed.
5. Patients with grade 2 CIPN with perceived improvement of symptoms.
6. Changes in neuropathic pain modulators will not be allowed.
7. Any other therapies for chemotherapy-induced peripheral neuropathy must be discontinued at least 2 weeks before the first dose of study drug.
8. Known hypersensitivity reaction to PSP Neuro serum.
9. Patients with a known or suspected shellfish allergy.
10. No dermatologic lesions on hands and feet and cuticles that might increase systemic exposure of the investigational medicinal product (IMP).
11. Distal muscle weakness and/or atrophy.
12. History of alcoholism or alcohol intake of 168g (21 units) for men and 112g (14 units) for women per week on a regular basis (time > 3 months). 1 unit = 10mL = 8g of pure alcohol.
13. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

    1. Diagnosis of type I or II diabetes mellitus (regardless of management) that have symptoms attributable to diabetic neuropathy pre-treatment with chemotherapy. Well-controlled diabetic patients (regardless of management), previously asymptomatic may be included.
    2. Glycosylated hemoglobin (HbA1C) ≥8.0% at screening.
    3. Fasting serum glucose ≥ 160 mg/dL at screening. Fasting is defined as no caloric intake for at least 8 hours.
14. Vitamin B12 deficiency defined as < 250 ng/mL.
15. Phosphate levels above upper limit of normal (ULN).
16. ECG: QTc interval (Fridericia Formula) ≥ 450ms.
17. Positive Tinel and/or Phalen test.
18. Participation in another clinical trial and any concurrent treatment with any investigational drug within 4 weeks prior to trial entry / randomization.
19. Surgery, radiotherapy, or systemic therapy that in the investigators' opinion might interfere/ worsen symptoms and the evaluation of peripheral neuropathy within 2 weeks prior to trial entry /randomization.
20. Any other finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patients at high risk from treatment complications.
21. Unresolved clinically significant toxicity from prior therapy except for alopecia.
22. Failure to adhere to study treatment and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-07-11 (Estimated); Study Completion 2025-07-14 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in response caused by PSP NEURO SERUM on the tactile sensation from baseline to day 28. | Screening and day 28
  The response will be assessed using the Semmes-Weinstein monofilament test.

SECONDARY OUTCOMES:
Evaluate the change in the overall neurological examination using the Total Neuropathy Score (TNSc), from baseline to day 28. | Screening and day 28.
  Evaluate the improvement of overall neurological examination as assessed by the clinical version of the Total Neuropathy Score (TNSc). The examination includes sensory symptoms, motors symptoms, autonomic symptoms, pin sensation, vibration sensibility, strength and tendon reflexes. The scores for each measurement goes from 0 to 4, being 0 a normal result and 4 an abnormal one.
Evaluate the change of manipulative dexterity and agility from baseline to day 28. | Screening and day 28.
  Evaluate the improvement of manipulative dexterity and agility as assessed through the NHPT (Nine-hole Pegboard Test - test of nine pins and holes).
Evaluate the change in patient reported symptoms from baseline to day 28. | Screening and day 28.
  Evaluate the improvement in patient reported symptoms as assessed by the EORTC CIPN20
Evaluate the appearance of Adverse Events according to NCI-CTCAE v5.0 (National Cancer Institute - Commun Toxicity Criteria For Adverse Events). | Through the 28 days of the study
  Evaluate safety and toxicity (type, frequency, grade and causality of adverse effects) of PSP NEURO SERUM according to NCI-CTCAE v5.0.
Evaluate the change in the quality of life from baseline to day 28. | Screening and day 28
  Evaluate the improvement of quality of life by using the Portuguese version of the 30-item European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) version.

CONTACTS AND LOCATIONS:
Overall Officials: Mariane Fontes, MD, Principal Investigator — Oncoclínicas
Locations (9):
- Brazil (9):
  - Oncoclínicas Vitória, Vitória, Espírito Santo
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Oncoclinicas do Brasil Servicios Medicos SA, Belo Horizonte, Minas Gerais
  - Centro Oncológico do Triângulo S.A., Uberlândia, Minas Gerais
  - Oncoclínicas João Pessoa, João Pessoa, Paraíba
  - Multihemo, Recife, Pernambuco
  - Oncoclínicas Florianópolis, Florianópolis, Santa Catarina
  - Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Centro de Paulista de Oncologia, São Paulo

IPD SHARING:
Plan to Share IPD: No